CLINICAL TRIAL: NCT04297553
Title: Outcomes of Fresh Transfer Versus Freeze-only After CAPA IVM on PCOS Patients
Brief Title: Fresh Versus Freeze-only After CAPA IVM on PCOS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS/BVMĐPN/20/01
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: PCOS; IVM; Embryo Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAPA-Fresh (Active Comparator): Receiving FSH (Menopur, Ferring) for 2 days on day 2/3 of the menstrual cycle (spontaneous/ OCP administration) and an ultrasound scan will be performed subsequently. Oocytes retrieval will be performed 42 hours after the last injection. Receiving hCG 5000IU x 2 (10000IU) after Oocytes retrieval. Pre-maturation will last for 24-30 hours. ICSI will be used for insemination. Fresh embryos transfer will be performed on day 3 using HRT protocol with a maximum of 2 embryos transferred.
  Interventions: Procedure: CAPA-Fresh
- CAPA-Freeze-only (Active Comparator): Receiving FSH (Menopur, Ferring) for 2 days on day 2/3 of the menstrual cycle (spontaneous/ OCP administration) and an ultrasound scan will be performed subsequently. Oocytes retrieval will be performed 42 hours after the last injection. Pre-maturation will last for 24-30 hours. ICSI will be used for insemination. Freeze-only on day 3 and frozen embryo transfer will be performed on the subsequent cycle using HRT protocol with a maximum of 2 embryos transferred
  Interventions: Procedure: CAPA-Freeze-only

INTERVENTIONS:
Procedure: CAPA-Fresh — Receiving FSH (Menopur, Ferring) for 2 days on day 2/3 of the menstrual cycle (spontaneous/ OCP administration) and an ultrasound scan will be performed subsequently. Oocytes retrieval will be performed 42 hours after the last injection. Receiving hCG 5000IU x 2 (10000IU) after Oocytes retrieval. Pre-maturation will last for 24-30 hours. ICSI will be used for insemination. Fresh embryos transfer will be performed on day 3 using HRT protocol with a maximum of 2 embryos transferred.
  Arms: CAPA-Fresh
Procedure: CAPA-Freeze-only — Receiving FSH (Menopur, Ferring) for 2 days on day 2/3 of the menstrual cycle (spontaneous/ OCP administration) and an ultrasound scan will be performed subsequently. Oocytes retrieval will be performed 42 hours after the last injection. Pre-maturation will last for 24-30 hours. ICSI will be used for insemination. Freeze-only on day 3 and frozen embryo transfer will be performed on the subsequent cycle using HRT protocol with a maximum of 2 embryos transferred.
  Arms: CAPA-Freeze-only

SUMMARY:
IVM (in vitro maturation) has been proved to be a more friendly treatment protocol for PCOS (polycystic ovary syndrome) patients compared with conventional controlled ovarian stimulation, with less complications (especially ovarian hyperstimulation syndrome), shorter treatment duration, lower cost, and acceptable pregnancy outcomes.

DETAILED DESCRIPTION:
IVM (in vitro maturation) has been proved to be a more friendly treatment protocol for PCOS (polycystic ovary syndrome) patients compared with conventional controlled ovarian stimulation, with less complications (especially ovarian hyperstimulation syndrome), shorter treatment duration, lower cost, and acceptable pregnancy outcomes. CAPA (capacitation) IVM without hCG (human chorionic gonadotropin) priming, has routinely been used at My Duc hospital for nearly 3 years to replace hCG-IVM (with hCG priming) because of absolutely synchronized oocyte maturation stage and better embryo results and better pregnancy outcomes. However, with CAPA IVM, embryos are freezed-only and will be transferred in the next cycles. This process will increase the cost of freezing and thawing embryos, and increase the treatment duration, which complicates the IVM procedure and turns IVM into an unfriendly protocol to PCOS patients. Therefore, our group conducts this study to find out the effectiveness of fresh transfer protocol after CAPA IVM compared with freezing-only CAPA IVM protocol. The fresh transfer protocol for CAPA IVM is applied from previous hCG IVM protocol, with the use of hCG and exogenous estradiol and progesterone, but at different timings.

ELIGIBILITY:
Inclusion Criteria:

* Women with high AFC (≥24 Antral Follicles in Both Ovaries), including PCOS plus PCO or high AFC
* Having indications for ART
* Having ≤ 2 IVM/IVF attempts
* Permanent resident in Vietnam
* Agree to have fresh embryos transfer or freeze-only on day 3
* Agree to have ≤ 2 embryos transferred
* Not participating in another IVF study at the same time

Exclusion Criteria:

* Oocyte donation cycles
* Pre-implantation genetic diagnosis (PGD) cycles

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy resulting in live birth after the first embryo transfer of the started treatment cycle. | At 24 weeks of gestation
  Live birth is defined as the birth of at least one newborn after 24 weeks' gestation that exhibits any sign of life (twin will be a single count).
  For the timing of this occur, ongoing pregnancy will be used, conditional on the fact that this ongoing pregnancy results in live birth.

SECONDARY OUTCOMES:
Positive pregnancy test | at 2 weeks after the embryo placement after the completion of the first transfer
  Serum human chorionic gonadotropin level greater than 5 mIU/mL
Clinical pregnancy | 5 weeks after embryo placement after the completion of the first transfer
  at least one gestational sac on ultrasound at 7 weeks' gestation with the detection of heart beat activity
Implantation rate | 3 weeks after embryo transferred after the completion of the first transfer
  as the number of gestational sacs per number of embryos transferred
Ongoing pregnancy | At 12 weeks' gestation
  Ongoing pregnancy is defined as pregnancy with detectable heart rate at 12 weeks' gestation or beyond, after the completion of the first transfer
Number of embryos on day 3 | 5 days after oocytes pick-up
  Number of embryos on day 3
Number of good quality embryo on day 3 | 5 days after oocytes pick-up
  good quality embryos are defined followed Istanbul consensus
Time from randomisation to ongoing pregnancy | 12 weeks of gestation after the completion of the first transfer
  Time from randomization to ongoing pregnancy after the completion
Time from randomisation to live birth | At the time of delivery
  Time from randomization to live birth after the completion
Ovarian hyperstimulation syndrome (OHSS) | at 03 days after oocytes pick-up and 14 days after embryo transfer
  Routine assessments for OHSS were performed on day 3 post oocyte retrieval in both groups. At other times, OHSS was evaluated if symptoms were reported by the patient. OHSS was classified using the flow diagram developed by Humaidan and colleagues for use in clinical trial settings
Ectopic pregnancy | at 12 weeks of gestation after the completion of the first transfer
  a pregnancy in which implantation takes place outside the uterine cavity after the completion of the first transfer
Miscarriage | at 24 weeks of gestation after the completion of the first transfer
  pregnancy loss at < 24 weeks
Hypertensive disorders of pregnancy | at 20 weeks of gestation or beyond after the completion of the first transfer
  Pregnancy-induced hypertension, pre-eclampsia and eclampsia
Gestational diabetes mellitus | at 24 weeks of gestation after the completion of the first transfer
  using a 75g oral glucose tolerance test
Preterm delivery | at 24, 28, 32 weeks and 37 weeks of gestation after the completion of the first transfer
  Multiple definitions, defined as delivery at <24, <28, <32, <37 completed weeks
Multiple pregnancy | 5 weeks after embryo placement after the completion of the first transfer
  Defined as presence of more than one sac at early pregnancy ultrasound (6-8 weeks gestation)
Birth weight | at the time of delivery
  Weight of singletons and twins
Congenital anomaly | At birth after the completion of the first transfer
  Any congenital anomaly will be included
Cost-effectiveness | Two year after randomization
  Including direct and indirect costs; costs related to complications treatment. Cost data will be collected for a supplementary analysis and will be reported in a separated paper.

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, MD, PhD, Principal Investigator — Mỹ Đức Hospital
Locations (1):
- Mỹ Đức Hospital, Ho Chi Minh City, Tan Binh, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vuong LN, Nguyen LK, Le AH, Pham HH, Ho VN, Le HL, Pham TD, Dang VQ, Phung TH, Smitz J, Ho TM. Fresh embryo transfer versus freeze-only after in vitro maturation with a pre-maturation step in women with high antral follicle count: a randomized controlled pilot study. J Assist Reprod Genet. 2021 Jun;38(6):1293-1302. doi: 10.1007/s10815-021-02180-7. Epub 2021 Apr 6. PMID 33825118